CLINICAL TRIAL: NCT01248299
Title: A Multicenter Randomized Phase II Study to Evaluate the Benefit of Chemotherapy Plus Best Supportive Care (BSC) Versus BSC in Patients With Metastatic Oesophageal Cancer of Squamous Cell-type Who Have Not Experienced a Disease Progression or Unacceptable Toxicity After a 6-weeks Chemotherapy Course .
Brief Title: Benefit of Chemotherapy Over Best Supportive Care in Metastatic and Squamous Cell-type Esophageal Cancer.
Acronym: E-DIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-DIS 2010-06; 2010-021439-16 (Other: IDRCB Number - AFSSAPS)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Squamous Cell Carcinoma of Esophagus
Keywords: Chemotherapy; Best Supportive Care
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 5-FU-CDDP protocol; Folfox protocol; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy plus best supportive care (Experimental): Chemotherapy plus best supportive care with follow up at each cycle of the treatment with FU-CDDP; LV5FU2-CDDP; FOLFOX; TPF
  Interventions: Drug: FU-CDDP; Drug: LV5FU2-CDDP; Drug: FOLFOX; Drug: TPF
- Best supportive care (Active Comparator): Best supportive care with follow up every 6 weeks
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: FU-CDDP — every 21 days:
  * Fluoro-uracil [800 mg/m2, day 1 to day 5]
  * CisPlatin [75 mg/m2, day 1 or day 2]
  Other Names: Fluoro-uracil+CisPlatin
  Arms: Chemotherapy plus best supportive care
Drug: LV5FU2-CDDP — every 14 days:
  * Elvorin [200 mg/m2, 2h IV, day 1 and day 2]
  * Fluoro-uracil [400 mg/m2 as a bolus, day 1 and day 2]
  * Fluoro-uracil [600 mg/m2, 22h continous infusion, day 1 and day 2]
  * CisPlatin [50 mg/m2, day 2]
  Other Names: Elvorin+Fluoro-uracil+CisPlatin
  Arms: Chemotherapy plus best supportive care
Drug: FOLFOX — every 14 days:
  * Oxaliplatin [85 mg/m2 by 2h infusion, day 1]
  * Fluoro-uracil [400 mg/m2 as a bolus, day 1 and day 2]
  * Fluoro-uracil [600 mg/m2, by 22h continous infusion, day 1 and day 2]
  * Elvorin [500 mg/m2, day 1 and day 2]
  Other Names: Oxaliplatin+Fluoro-uracil+Elvorin
  Arms: Chemotherapy plus best supportive care
Drug: TPF — every 21 days:
  * Docetaxel [30 mg/m2, day 1 and day 8]
  * CisPlatin [60 mg/m2, day 1]
  * Fluoro-uracil [200 mg/m2/day by continous infusion]
  Or every 21 days:
  * Docetaxel [50 mg/m2, day 1]
  * CisPlatine [70 mg/m2, day 1]
  * Fluoro-uracile [700 mg/m2 /day, day 1 to day 5]
  Other Names: Docetaxel+CisPlatine+Fluoro-uracile
  Arms: Chemotherapy plus best supportive care
Other: Best Supportive Care — See European professionnal recommendations (ESMO 2009) Exemples : antalgic treatment, nutritional support, ...
  Other Names: antalgic treatment, nutritional support, ...
  Arms: Best supportive care

SUMMARY:
Interest of continuing systemic chemotherapy or not , after a short initial treatment (6 weeks) in patients who are in response or stable disease("Discontinuation design ")of patients with metastatic oesophageal cancer of squamous cell type

The secondary aims would be to study : toxicity, the overall survival rate, a study of costs and quality of life.

DETAILED DESCRIPTION:
As the data in litterature does not provide the basis for well-argued statistical hypothesis, it is suggested to randomize 30 patients per arm. An IDMC will come to a decision after the inclusion of 10, 20 ans 40 patients on the efficacy and the toxicity profile and on whether to maintain the current clinical position, justifying randomisation . In order to take into account any possible effects of prior concomitant radiochemotherapy, patient will be stratified according to whether they have already undergone chemotherapy or radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an histologically proven epidermoid cancer of the oesophagus
* Patients with metastatic disease that can be measured or evaluated according to the RECIST criteria, and located outside of previously irradiated fields
* Patients who may or may not have undergone radiochemotherapy
* Patients who have not received chemotherapy for metastatic disease
* ≥ 18 ans
* Performance Status (ECOG) ≤ 2
* People who are covered by private or state health insurance
* Informed consent signed by the patient

Exclusion Criteria:

* Other evolutive malignant tumor
* Infection with HIV-1, HIV-2 or chronic hepatitis B or C
* Cerebral metastasis or known meningeal tumor
* Any unstable chronic diseases that could risk the safety or the compliance of te patient
* Women who are pregnant or breastfeeding. Women must not breastfeed for at least 6 months after administration of Bevacizumab
* Patients unable to undergo the follow-up of the trial for geographical, social or psychological reasons

For the randomized part

Inclusion criteria :

* Non-progressive disease after the 6 first weeks of chemotherapy
* Performance Status (ECOG) ≤ 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Between the date of randomisation and the date of death

SECONDARY OUTCOMES:
Progression free survival | Between the date of randomisation and the date of progression
Tolerance | At each visit : every 6 weeks
  According to the NCI-CTCAE V4.0 grading scale
Quality of life by QLQ-C30 | Every 6 weeks
  EOTRC QLQ-C30 questionnaire and the oesophagus QLQ-OES18 module
  EQ-5D questionnaire
Cost analysis | Every 6 weeks
  Data collected :
  * Hospitalization
  * day hospital visit
  * Chemotherapy drugs administered
  * Home medical care
  * Radiotherapy
  * Oncologist visits, General Practitioner Visits
  * Laboratory and radiologic tests

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (17):
- France (17):
  - CHU Brest, Brest
  - Centre François BACLESSE, Caen
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - Centre Oscar Lambret, Lille
  - CHU Lille, Lille
  - CHU La Timone, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Eugène Marquis, Rennes
  - Clinique de la Theuillerie, Ris-Orangis
  - CHU Rouen, Rouen
  - Clinique de l'Armoricaine, Saint-Brieuc
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecki N, Hiret S, Etienne PL, Penel N, Tresch E, Francois E, Galais MP, Ben Abdelghani M, Michel P, Dahan L, Ghiringelli F, Bedenne L, Samalin E, Piessen G, Bennouna J, Peugniez C, El Hajbi F, Clisant S, Kramar A, Mariette C, Adenis A. First-Line Chemotherapy for Metastatic Esophageal Squamous Cell Carcinoma: Clinico-Biological Predictors of Disease Control. Oncology. 2016;90(2):88-96. doi: 10.1159/000442947. Epub 2016 Jan 20. PMID 26784946